CLINICAL TRIAL: NCT02852759
Title: A Cold Physical Treatment to Manage Insulin Resistance
Acronym: CTPMIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF-CRS-2016-018
Record Dates: First submitted 2016-07-20; First posted 2016-08-02 (Estimated); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Insulin Resistance; Hyperglycemia; Hyperinsulinemia; Diabetes; Obesity
MeSH Terms: conditions — Insulin Resistance; Hyperglycemia; Hyperinsulinism; Diabetes Mellitus; Obesity | interventions — Electroacupuncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention group (Experimental): Add Selective Cold and Electroacupuncture treatment to the existing treatment for patients with insulin resistance.
  Interventions: Procedure: Selective Cold; Device: Electroacupuncture
- Intensive Care group (No Intervention): continue the existing management of insulin resistance in these patients. They will receive the same follow up, examinations etc as intervention group.

INTERVENTIONS:
Procedure: Selective Cold — The volunteers of intervention group will undergo Selective Cold treatment below 10 degree celsius to neck, supraclavicular interscapular regions for 2 hours daily for 8 weeks. The electroacupuncture is conducted by commercially available device. Hyperinsulinemic euglycemic clamp, glucose tolerance test, blood parameter measurements, and PTC-CT scans will be conducted before and after the intervention. The participants will be instructed to maintain their normal behavior and calorie intake.
  Arms: intervention group
Device: Electroacupuncture — Electroacupuncture (EA) is an add-on treatment and it is applied when starting the cold treatment at the cold treated region to patients.The device is Huatuo SDZ-II model made by Suzhou Medical Appliance Factory, China.
  Arms: intervention group

SUMMARY:
Insulin resistant volunteers will choose to undergo an 8-week cold treatment, 2 hours per day, to selective regions of the body enriched with brown fat including neck, supraclavicular and interscapular regions) in combination with electroacupuncture (EA). Their insulin sensitivity and glucose and lipid homeostasis will be measured. The brown fat activation will be assessed by positron emission tomography and computed tomography (PET/CT)-scans and/or serum marker measurements.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 20-30
* Insulin resistant

Exclusion Criteria:

* uncontrolled hypertension
* insulin dependent diabetics
* heart diseases
* hyperthyroidism
* secondary obesity
* surgical operation within treatment or planned in two months
* pregnancy
* anemia
* liver or kidney failure
* cancer

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Change of Glucose Tolerance measured by OGTT | 0, 8 week, 2 hours for each measurement
  glucose tolerance at 8 weeks will be compared to 0 week

SECONDARY OUTCOMES:
Change of serum insulin levels | 0, 8 week
  8 weeks will be compared to 0 week
Change of Body weight | 0, 8 week
  8 weeks will be compared to 0 week
Change of 2-deoxy-2-[fluorine-18]fluoro- D-glucose (FDG) uptake by PET/CT-scans | 0 and 8 week, 2 hours for each measurement
  8 week will be compared to 0 week
Change of glucose infusion rate by hyperinsulinemic euglycemic clamp | 0 and 8 week, 5 hours for each measurement
  8 week will be compared to 0 week

CONTACTS AND LOCATIONS:
Overall Officials: Li Qiang, Ph.D., Principal Investigator — Columbia University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: Yes
Study result will be published after finishing the trial